CLINICAL TRIAL: NCT05343754
Title: Hyperbaric Oxygen Therapy for Pyoderma Gangrenosum As a New Treatment Strategy
Brief Title: Hyperbaric Oxygen Therapy for Pyoderma Gangrenosum
Acronym: HOTPANTS
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Due to low recruitment
Sponsor: Erasmus Medical Center (Other)
Responsible Party: Principal Investigator, K.R. van Straalen, Pincipal investigator, Erasmus Medical Center
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: NL 2021-006013-11
Record Dates: First submitted 2022-04-11; First posted 2022-04-25 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2022-07

CONDITIONS: Pyoderma Gangrenosum
Keywords: Hyperbaric Oxygen Therapy
MeSH Terms: conditions — Pyoderma Gangrenosum | interventions — Hyperbaric Oxygenation; Respiration; Control Groups

STUDY DESIGN:
Intervention Model Description: The study design is a pragmatic prospective cohort study: a group of patients with therapy refractory pyoderma gangrenosum despite standard wound care and anti-inflammatory treatment for at least 6 weeks will be treated with hyperbaric oxygen therapy.
Masking Description: Patients are aware of another treatment possibility (hyperbaric Oxygen therapy) which will be investigated.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Hyperbaric Oxygen Therapy (Active Comparator): Hyperbaric treatment will consist of 30 daily treatments in the first 6 weeks of the study, except during the weekends. After compression for 10 minutes patients will receive 80 minutes (4 times 20 minutes) 100% O2 with 3 airbrakes (21% O2) of 5 minutes at 2.4-2.5 ATA, and then 10 minutes decompression with the first part of decompression till 0.3 ATA with 100% oxygen (this will usually take seven minutes). The last 0.3 ATA will be decompressed with air. In total one hyperbaric session will be 110 minutes. Treatment will start directly at the beginning of the study.
  Interventions: Drug: Hyperbaric oxygen
- Control group (Active Comparator): In order to compare efficacy, patients that do not wish to undergo hyperbaric treatment, will serve as a control group. At baseline they will be asked for the reason they do not wish to undergo hyperbaric treatment. All patients and controls will be asked to report pain scores using a numeric pain rating scale (NRS) and quality of life (Wound-Q) questionnaires. They will continue to receive standard care as deemed necessary by their primary physician.
  Interventions: Other: Control group

INTERVENTIONS:
Drug: Hyperbaric oxygen — Hyperbaric treatment will consist of 30 daily treatments in the first 6 weeks of the study, except during the weekends. After compression for 10 minutes patients will receive 80minutes (4 times 20 minutes) 100% O2 with 3 airbrakes (21% O2) of 5 minutes at 2.4-2.5 ATA, and then 10 minutes decompression with the first part of decompression till 0.3 ATA with 100% oxygen (this will usually take seven minutes). The last 0.3 ATA will be decompressed with air. In total one hyperbaric session will be 110 minutes. Treatment will start directly at the beginning of the study.
  Other Names: breathing 100% oxygen under hyperbaric circumstances
  Arms: Hyperbaric Oxygen Therapy
Other: Control group — In order to compare efficacy, patients that do not wish to undergo hyperbaric treatment, will serve as a control group. At baseline they will be asked for the reason they do not wish to undergo hyperbaric treatment. All patients and controls will be asked to report pain scores using a numeric pain rating scale (NRS) and quality of life (Wound-Q) questionnaires. They will continue to receive standard care as deemed necessary by their primary physician.
  Other Names: standard wound care
  Arms: Control group

SUMMARY:
Rationale: Pyoderma gangrenosum (PG) is a rare auto-inflammatory neutrophilic dermatosis characterized by a spectrum of clinical presentations with variable courses. Diagnosis and management are challenging in PG. Treatment, including systemic prednisone and anti-TNF therapy, is directed towards reducing pain and associated inflammation that leads to ulceration. Positive effects of hyperbaric oxygen (HBO) therapy have been reported in small case series.

Objective: To investigate the therapeutic efficacy of hyperbaric oxygen on top of standard wound care and regular anti-inflammatory treatment in patients with pyoderma gangrenosum wounds.

Study design: Prospective cohort study with a follow-up to one year. Study population: 15 adult patients with pyoderma gangrenosum refractory to standard-prednisone or anti-TNF therapy will be included for hyperbaric oxygen therapy. Patients with pyoderma gangrenosum that are eligible but reject hyperbaric oxygen treatment will serve as controls. In total the investigators will include 30 patients.

Intervention (if applicable): 30 sessions of HBO therapy will be applied on top of regular wound care and systemic anti-inflammatory treatment. Controls will be treated with regular wound care and anti-inflammatory treatment.

Main study parameters/endpoints: Wound healing time (time to wound closure). PG wounds will be measured at baseline using a validated, objective 3D photographical wound measurement tool, and again after 3 and 6 weeks at the end of HBO treatment and after 3 months. Patients will take weekly photographs at home using a 2D validated measurement tool of the wounds.

Secondary parameters: Alteration in the expression of markers of inflammation by micro-biopsies of wound edges, non-invasive mitochondrial O2 measurements at wound edges, blood neutrophil count and patient-reported outcomes like WOUND-Q, pain on NR scale and treatment satisfaction scores. Assessment concerning laboratory findings will be done at baseline before starting the trial, at 3 weeks and at week 6 at the end of HBO treatment. Patient reported outcomes, WOUND-Q will be measured at baseline, 3 weeks, 6 weeks, 3 months, 6 months, and 12 months. Mean NRS scores will be recorded once a week.

DETAILED DESCRIPTION:
INTRODUCTION AND RATIONALE

Pyoderma gangrenosum (PG)

Background information Pyoderma gangrenosum (PG) is a rare, uncommon auto-inflammatory neutrophilic dermatosis characterized by a spectrum of clinical presentations including painful chronic and recurrent cutaneous ulcers with a necrolytic border with variable courses. PG has an overall prevalence of 5 to 10 per 100,000 individuals and an increased mortality rate compared with the general population. Its pathophysiology is complex and not fully understood. PG affects patients of both sexes equally and of any age, although female predominance has also been reported, with a peak incidence between 20 and 50 years of age. Legs are most commonly affected but head, trunk and neck involvement are not uncommon in children, while involvement of the genital and perianal area has been reported in adults as well in infants. There are multiple subtypes of PG, including ulcerative (A), bullous (B), pustular (C), vegetative (D) (pyostomatitis vegetans), peristomal, drug-induced and post-surgical PG (E).

Pathergy, an exaggeration of skin injury occurring after minor trauma, is seen in one-third of patients with PG and can contribute to peristomal and post-surgical PG (PSPG). PSPG occurs at the site of surgery, most commonly reported after breast, chest, or cardiothoracic surgery. PG is considered a "diagnosis of exclusion of clinical features" due to lack of definitive laboratory or histopathological diagnostic criteria and is thus frequently misdiagnosed.

Pathophysiology The pathophysiology of PG represents a complex inflammatory reaction pattern with involvement of multiple pathways that results in a heterogeneous disease presentation and course. The course of PG can vary from relatively indolent to aggressive or fulminant to fatal. Involvement of innate and adaptive immune dysregulation, genetic variants, as well as neutrophilic abnormalities have been described. PG is associated with other neutrophilic or inflammatory disorders such as inflammatory bowel disease (both Crohn's disease and Colitis Ulcerosa), rheumatoid arthritis, suppurative hidradenitis, seronegative arthritis, autoimmune hepatitis, and hematologic disorders, including paraproteinemia, especially IgA, and (neutrophilic) malignancies such as acute and chronic myelogenous leukemia. There are also associations with rare genetic disorders with pyoderma gangrenosum respectively Pyogenic Arthritis Pyoderma Acne (PAPA), Pyoderma Acne Suppurative Hidradenitis (PASH), Pyogenic Arthritis Pyoderma Acne Suppurative hidradenitis (PAPASH), and Pyoderma Acne ulcerative Colitis (PAC).3,7-10 Elevated levels of inflammatory mediators have been found in lesions of PG, suggesting a pathological inflammatory process. PG lesions show significant overexpression of cytokines like IL-1α, IL-1β, IL-6, IL-8, IL-12, IL-17, IL-23, IL-36α, TNF, matrix metalloproteinases, endothelial- and leukocyte-selectins. In the adaptive system the ratio between T regulatory cells and Th17 cells was found to be reduced in PG lesions. There are still several unknown factors, including the initiating trigger for immune dysregulation as well as additional contributory components of the immune system.

Diagnosis Separate diagnostic tools for PG have been published, among others by Su et al in 2004, Maverakis et al in 2018 and by Jockenhöfer in 2019. These tools include major and minor criteria for the probability of the diagnosis of PG. Biopsy, cultures, blood tests such as testing for ANCA's and more are necessary to exclude other diagnosis or in particular underlying not yet diagnosed related diseases. PG is challenging to both diagnosis and management, and treatment is directed towards reducing the associated inflammation that leads to ulceration. In this prospective pragmatic trial, both the PARACELSUS as well as the Delphi criteria will be used to confirm the diagnosis of pyoderma gangrenosum (Appendix 1. PARACELSUS acronym and criteria

Treatment The choice of treatment depends on numerous factors, including location of lesion(s), number, size, extra cutaneous involvement, presence of associated diseases, aggressiveness of the disease, costs or reimbursement possibilities, and side effects of treatment, as well as patient comorbidities and preferences. Treatment includes general measures lifestyle changes, advanced wound care, topical therapy such as potent topical corticosteroids, systemic therapy with corticosteroids and targeted therapy like anti-TNF, anti-IL-1 or anti-IL-12/23 (Figure 3 and 4).The mean wound healing time in patients treated with anti-TNF biologics is 86,1 days, compared with a mean wound healing time of 168 days in 47% of patients treated with cyclosporine or prednisolone.

Hyperbaric oxygen therapy Hyperbaric oxygen therapy is a safe treatment procedure that involves breathing 100% oxygen under higher-than-normal atmospheric pressure, usually 2.0-2.5 atmosphere absolute (ATA). Delivering 100% oxygen to the lungs leads to an increased level of plasma and tissue oxygen levels and decreases hypoxia. HBOT is commonly used in the treatment of decompression sickness, carbon monoxide intoxication, arterial gas embolism, necrotizing soft tissue infections, late radiation injury with or without chronic wounds, diabetic (foot) ulcers and severe multiple traumata with ischemia. Figure 5 is an example of standard hyperbaric treatment given in multiplace centers in The Netherlands. After compression for 10 minutes patients will receive 75 minutes (4 times 20 minutes) 100% O2 with 3 airbrakes (21% O2) of 5 minutes at 2.4-2.5 ATA, and then 10 minutes decompression with the first part of decompression till 0.3 ATA with 100% oxygen, which will usually take seven minutes. The last 0.3 ATA will be decompressed with air. In total one hyperbaric session will last 110 minutes.

HBOT mechanisms The increased level of plasma and tissue oxygen levels with HBOT is valuable for the healing of inflammatory and microcirculatory disorders in ischemic circumstances and the compartment syndrome. HBO has been shown to alter signaling pathways such as Hypoxia Induced Factor (HIF) and heme-oxygenase (HO), both involved in issue response to hypoxia and wound repair.21-23 Also, in general, oxidative stress is recognized to play a role in stem cell mobilization and to promote wound healing. HBOT enhances (neo-)angiogenesis and cell proliferation, which results in the formation of granulation tissue and subsequent improvement of wound healing.

The anti-inflammatory effects of HBOT have been reported to play a key role in reducing tissue damage and infection development. HBOT induces overexpression of growth factors and down-regulation of pro-inflammatory cytokines to subsequently reduce immune responses. The increased oxygen levels during HBOT is demonstrated to cause cellular effects such as the suppression of various cytokines like interferon-gamma, pro-inflammatory cytokines such as IL-1, IL-6, and TNF, a transient decrease in the CD4:CD8 T cell ratio, the reduction of serum soluble IL-2 receptor (sIL-2R) levels, enhancement of plasma fibronectin , significant elevation of IL-10, inhibition of TGFβ-pathway and induction of lymphocyte apoptosis by a mitochondrial pathway. In short, HBOT induces an anti-inflammatory program across several pathways.

Rationale Standard advanced wound care in pyoderma gangrenosum consists of topical and systemic treatments. Aggressive surgical debridement in pyoderma gangrenosum should be avoided, because of high risk of wound aggravation. The aforementioned combined therapies are described in case reports with or without adjuvant HBOT. Barr et al. was the first in 1972 to report the successful treatment of pyoderma gangrenosum with HBOT. In several other case reports additional HBOT yielded excellent responses in cases of refractory pyoderma gangrenosum. Mean number of sessions of HBOT needed before remission were respectively 29 and 31 in total, with a range from 11 to 86. Because Pyoderma gangrenosum is an auto-inflammatory disease and mostly associated with other auto inflammatory disorders like rheumatoid arthritis and Inflammatory Bowel Disease (both Colitis ulcerosa and M. Crohn), case reports and series show a good response with adjunctive HBOT with a mean wound healing time of 40,25 days (5,75 weeks with a range of 10 to 90 days).

The anti-inflammatory mechanisms of HBOT at the cellular and cytokine levels in chronic ulcers are most likely the keystone of success of adjuvant HBO treatment of refractory pyoderma gangrenosum. Based on the mechanisms of HBOT mentioned above, like suppression of proinflammatory cytokines like TNF, IL-1, IL-6, reduction in MMPs, neutrophil activation as well reduction in T cell subsets, the investigators hypothesize that HBOT may have a positive effect on pyoderma gangrenosum. In addition to the clinical response, our proposed trial will assess in a prospective cohort the effects and the molecular mode of action of advanced wound care with and without HBOT on wound healing, pain and PROMs in pyoderma gangrenosum.

Hypothesis Based on several case reports a positive effect of HBOT on wound healing time is expected.

A significant shorter wound healing time with HBOT can reduce the necessary expensive use of hospitalization and third line medication like TNF inhibitors.

HBOT exerts an anti-inflammatory effect on local PG inflammation. Does HBOT prevent recurrence of PG?

OBJECTIVES

Primary objective To compare the clinical efficacy of HBO treatment on top of standard regular wound care and anti-inflammatory treatment in patients with PG, with time to wound closure as the primary outcome, using a validated, objective 2D and 3D photographical wound measurement tools. Controls will be treated with regular wound care and anti-inflammatory treatment.

Secondary objectives

* Changes in markers of inflammation, mRNA expression in micro-biopsies in wound edges.
* Alterations in mitochondrial O2 levels
* The number of activated neutrophils in peripheral venous blood.
* To assess the effect of HBOT on Pain reduction (NRS score).
* To assess the effect of HBOT on Health Related-Quality of Life (WOUND-Q).
* To assess the prevalence of recurrence of PG in patients treated with and without adjuvant HBOT.

STUDY POPULATION Population (base) Inclusion of patients with a confirmed diagnosis of a pyoderma gangrenosum wound, refractory to standard wound care and anti-inflammatory systemic treatment. These patients will be recruited at the outpatient clinic of the dermatology, clinical immunology or rheumatology department in the Erasmus Medical Center Rotterdam and affiliated peripheral general hospitals. The planned number of 15 patients for hyperbaric treatment and 15 controls can be recruited from external clinics given the referral population that see 5-10 patients per year per dermatological department and referred to the ErasmusMC for further follow-up. Patients that wish to participate but turn down hyperbaric treatment will serve as a control group.

Inclusion criteria

In order to be eligible to participate in this study, a subject must meet all of the following criteria:

* Confirmed consensus on the diagnosis pyoderma gangrenosum by referring specialist, principal and coordinating investigator (dermatologist, clinical immunologist or rheumatologist based on PARACELSUS and Delphi score).
* Unsatisfactory response after six weeks of combined standard wound care and systemic prednisone and/or other anti-inflammatory therapy.
* Fit for hyperbaric oxygen therapy as assessed by the hyperbaric physician.
* Age ≥18 years at baseline
* All genders
* Able and willing to give written informed consent and to comply with the study requirements.

Exclusion criteria

A potential subject who meets any of the following criteria will be excluded from participation in this study:

* Language barrier
* Unable to give informed consent or to comply with the trial protocol
* Pregnancy

Sample size calculation The primary outcome is defined as the fraction of patients with complete wound healing at three months. Assuming that this is 0.2 in the control group and 0.7 in the experimental group. Fixing the test size at 0.05 the investigators need 15 patients in the HBOT group and 15 patients in the control group. In total the investigators need 30 subjects to achieve a power of 80%.

Investigational product/treatment Hyperbaric oxygen therapy: subjects will be placed in the hyperbaric chamber and breath room air or 100% oxygen through a non-rebreathing mask after the tank is pressurized to 2.4-2.5 ATA. The duration of this protocol (total of 80 minutes of breathing 100% oxygen with 5-minute breaks on normal air, total session time: 110 minutes). This HBOT-regimen is similar to the normal clinical HBO protocol in The Netherlands and thus remains well within non-decompression and oxygen toxicity limits. Patients allocated to the intervention group will receive 30 sessions of HBOT excluding the weekend adjunctive to standard care. In order not to interrupt the induction of anti-inflammatory and wound healing effects (which take place at the beginning of treatment): if patients for whatever reason miss more than 2 sessions in the first four weeks, the treatment regimen will be restarted from the beginning.

The hyperbaric treatment takes place in any of the following hyperbaric facilities if this will be closer for patients:

* Da Vinci Clinics Netherlands: Rotterdam, Waalwijk, Arnhem, Hoogeveen, Amersfoort or Geldrop
* Hyperbaric Medical Centre Rijswijk
* Medical Centre Hyperbaric Oxygen Therapy Goes
* Hyperbaric Centers Belgium

In this trial, oxygen will be used under hyperbaric conditions. In addition, 100% oxygen will be administered. Both can be either cryogenic preserved oxygen or compressed oxygen.

Summary of findings from non-clinical studies For the scope of this study the finding in non-clinical studies is not relevant, since HBOT is already widely implemented in humans and clinical studies are available.

Summary of findings from clinical studies HBOT has a variety of mechanisms of action: it improves tissue oxygenation; inhibits the pro-inflammatory reaction by reducing cytokines; improves neo-vascularization; has a bacteriostatic effect on anaerobic bacteria and stimulates stem cells and growth factors. There are 14 indications of HBOT approved by the UHMS, including the treatment of air or gas embolism, arterial insufficiencies, carbon monoxide poisoning and gas gangrene.

A deeper understanding of the role of oxygen was provided by Kaelin, Ratcliffe and Semenza, who discovered how cells can sense and adapt to changing oxygen availability (for which they received the Nobel Prize of Physiology or Medicine in 2019). They identified molecular machinery that regulates the activity of genes in response to varying levels of oxygen.

Summary of known and potential risks and benefits

Risks: HBOT might cause middle ear and sinus barotrauma, myopia, and epileptic seizures; see the structured risk analysis.

Benefits: patients could potentially benefit from this treatment in terms of faster wound healing time, pain reduction, improved health and quality of life.

Description and justification of route of administration and dosage Hyperbaric treatment will consist of 30 daily treatments (6 weeks, excluding the weekends), breathing 100% oxygen at a pressure of 2.4 - 2.5 atmosphere absolute (ATA). Every 20 minutes an air brake will be implemented, where patients only breathe room air. The total duration of one treatment is 110 minutes. This reduces risks of oxygen toxicity.

Dosages, dosage modifications and method of administration Depending on local protocols, patients will breathe 110 minutes of HBOT under 2.4-2.5 ATA. The total number of sessions will be 30.

6.7 Preparation and labelling of Investigational Medicinal Product All centers have to record the quality certificates of the oxygen used for patients included in the trial.

Drug accountability The shipment, receipt, disposition, return and destruction of oxygen will not be affected by this study. All HBOT-centers already have to record the quality certificates of the oxygen used for patients included in the trial.

STATISTICAL ANALYSIS

All parameters will be assessed for a two-tailed significance of p < 0,05.

Primary study parameter(s) The primary endpoint of this trial is the time to wound closure which represents a (semi-) continuous variable and will be analyzed with the non-parametric Wilcoxon signed rank test. Differences in wound healing time between the HBO group and control group will be analyzed using the unpaired t-test or Mann-Whitney U test.

Secondary study parameter(s) Differences in (semi-)continuous variables before and after treatment, such as the patient-reported outcomes (NRS scores, WOUND-Q), cytokine-mRNA in wound biopsies, laboratory venous blood findings (neutrophils, leucocytes and CRP), will be analyzed with the non-parametric Wilcoxon signed rank test. For differences between the HBO group and the control group the unpaired t-test or Mann-Whitney U test will be used.

Other study parameters Patient characteristics and demographic data as measured at baseline will be presented with continuous data as mean ± SD and categorical data as number (%), and analyzed using descriptive statistics. Differences in baseline characteristics between groups (intervention and control) will be assessed and included in the interpretation of results.

Interim analysis No interim analysis will be done.

ELIGIBILITY:
Inclusion Criteria:

* - Confirmed consensus on the diagnosis pyoderma gangrenosum by referring specialist, principal and coordinating investigator (dermatologist, clinical immunologist or rheumatologist based on PARACELSUS and Delphi score).
* Unsatisfactory response after six weeks of combined standard wound care and systemic prednisone and/or other anti-inflammatory therapy.
* Fit for hyperbaric oxygen therapy as assessed by the hyperbaric physician.
* Age ≥18 years at baseline
* All genders
* Able and willing to give written informed consent and to comply with the study requirements.

Exclusion Criteria:

* - Language barrier
* Unable to give informed consent or to comply with the trial protocol
* Pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2022-06-01 (Actual); Primary Completion 2024-01-14 (Actual); Study Completion 2024-01-14 (Actual)

PRIMARY OUTCOMES:
Wound healing time | 3 months
  To compare the clinical efficacy of HBO treatment on top of standard regular wound care and anti-inflammatory treatment in patients with PG, with time to wound closure as the primary outcome, using a validated, objective 2D and 3D photographical wound measurement tools. Controls will be treated with regular wound care and anti-inflammatory treatment.

SECONDARY OUTCOMES:
Cytokines changes | 6 weeks
  mRNA expression of cytokines in micro-biopsies in wound edges.
mitochondrial O2 levels | 6 weeks
  Alterations in mitochondrial O2 levels
Neutrophil count in peripheral venous blood | 6 weeks
  The number of activated neutrophils in peripheral venous blood.
pain dairy | 3 months
  Weekly pain dairy questionnaires, with 10 as the worst outcome and zero as the best outcome.
quality of life measurement | 1 year
  wound quality of life questionnaire; higher scores will be a better outcome than lower scores in QOL.

CONTACTS AND LOCATIONS:
Overall Officials: Errol Prens, Prof.Dr., Principal Investigator — Erasmus MC, dermatology department
Locations (1):
- Erasmus MC, Rotterdam, Netherlands

IPD SHARING:
Plan to Share IPD: No